CLINICAL TRIAL: NCT00005102
Title: Immunologic Evaluation in Patients With DiGeorge Syndrome or Velocardiofacial Syndrome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: Children's Hospital of Philadelphia (Other)
Other Study IDs: NCRR-M01RR00240-1571; CHP-IRB-95-903; CHP-GCRC-1571
Record Dates: First submitted 2000-04-06; First posted 2000-04-07 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: DiGeorge Syndrome; Shprintzen Syndrome; Chromosome Abnormalities; Abnormalities, Multiple; Conotruncal Cardiac Defects
Keywords: DiGeorge syndrome; Shprintzen syndrome; cardiovascular and respiratory diseases; conotruncal cardiac defects; genetic diseases and dysmorphic syndromes; rare disease
MeSH Terms: conditions — DiGeorge Syndrome; Chromosome Aberrations; Abnormalities, Multiple; Conotruncal cardiac defects; Respiratory Tract Diseases; Genetic Diseases, Inborn; Rare Diseases

STUDY DESIGN:
Observational Model: Natural History

SUMMARY:
OBJECTIVES:

I. Determine the pattern of immunologic reconstitution in patients with T-cell compromise due to DiGeorge syndrome or velocardiofacial syndrome.

II. Determine any correlation between immunologic function in these patients and chromosome 22 deletion breakpoints.

III. Determine presence of sustained immunologic compromise in older patients.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE:

Blood samples are collected at diagnosis of chromosome 22q11 deletion and assessed for lymphocyte proliferation in response to mitogens phytohemagglutinin, pokeweed mitogen, and concanavalin A (mitogen stimulation analyses). These analyses are repeated at 4 months along with a quantitative analysis of immunoglobulin.

At 8 months, patients are tested for their lymphocytes' ability to respond to antigens (candida, tetanus, and diphtheria). At 1 year, patients have lymphocyte subset, IgG, IgA, and IgM analyses performed. Quantitative evaluations of antibody titers to diphtheria, tetanus, Haemophilus influenza, and hepatitis B are also performed.

Over 1 year of age, all studies are performed if the patient is seen for a single visit.

ELIGIBILITY:
* Conotruncal cardiac lesion to be repaired by surgery AND Chromosome 22q11 deletion by FISH

Min Age: 0 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 11
Dates: Start 1995-01

CONTACTS AND LOCATIONS:
Overall Officials: Kathleen E. Sullivan, Study Chair — Children's Hospital of Philadelphia
Locations (1):
- Children's Hospital of Philadelphia, Philadelphia, Pennsylvania, United States